CLINICAL TRIAL: NCT06876532
Title: Evaluation of the Inflammation-based Index as a Predictive Marker of Clinical and Radiological Response in Patients Treated With Lu-177 Oxodotreotide for Intestinal Neuroendocrine Tumour
Acronym: LUTIBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24DIGE02
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Intestinal Neuroendocrine Tumor
Keywords: Intestinal Neuroendocrine Tumor; Lu-177 oxodotreotide; IBI score; Biomarker
MeSH Terms: interventions — Serum Albumin; Data Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Treated With Lu-177 Oxodotreotide for Intestinal Neuroendocrine Tumour (Other)
  Interventions: Other: Additional blood tests (CRP and serum albumin) and data collection.

INTERVENTIONS:
Other: Additional blood tests (CRP and serum albumin) and data collection. — These blood tests will be carried out on several occasions (before, during and after treatment with Lu-177 oxodotreotide). No additional blood sampling is required.
  In addition, patient clinical data and imaging data (standard examinations: thoraco-abdomino-pelvic CT +/- MRI and Ga-68 DOTA PET-CT) will be specifically collected for study purposes.
  For IUCT-O patients only: blood samples may be taken (at cycles 1 and 2, then 12 months after inclusion) for bio-banking purposes.

SUMMARY:
This is a prospective, multicenter, open-label study designed to evaluate the specificity and sensitivity of the Inflammation Based Index (IBI) score as a marker for predicting clinical and radiological response in patients treated with Lu-177 oxodotreotide for inoperable or metastatic, progressive, grade 1 or 2 intestinal neuroendocrine tumors.

This IBI score will be assessed on the basis of C-reactive protein (CRP) and albumin values, and will be defined as follows:

* IBI = 0: Low mortality risk (if CRP and serum albumin values are considered normal in the investigator's judgment).
* IBI > 0, including: IBI = 1: Intermediate risk of mortality (if one of the two values is considered abnormal and clinically significant according to the investigator's judgment (either hypoalbuminemia or elevated CRP)); IBI = 2: High mortality risk (if both values are considered abnormal and clinically significant according to the investigator's judgment (hypoalbuminemia and elevated CRP)).

Patients were followed up for 36 months.

A total of 150 patients should be included in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 18 years.
2. Patient with histologically confirmed grade 1 or 2 neuroendocrine tumor of the midgut, inoperable or metastatic.
3. Patient eligible for Lu-177 oxodotreotide therapy in accordance with its marketing authorization.
4. Evidence of progression in the 12 months preceding Lu-177oxodotreotide therapy, confirmed by imaging techniques commonly used in current practice (thoraco-abdomino-pelvic CT and/or liver MRI, Ga-68 DOTA somatostatin analog PET-CT) +/- liver involvement greater than 50%.
5. Disease measurable according to RECIST 1.1 criteria in thoraco-abdomino-pelvic CT +/- liver MRI.
6. Patient affiliated to a social security scheme in France.
7. Patient having signed informed consent prior to study inclusion and prior to any specific study procedure.

Exclusion Criteria:

1. Previous treatment with Lu-177 oxodotreotide.
2. Any contraindication to treatment with Lu-177 oxodotreotide.
3. Morbid obesity (BMI > 40).
4. Uncontrolled/unbalanced active inflammatory disease in the 3 months prior to inclusion.
5. Active carcinoid heart disease or other acute cardiovascular event.
6. Active infection not treated within 15 days.
7. Pregnant or breast-feeding woman.
8. Any psychological, family, geographical or sociological condition that prevents compliance with the medical follow-up and/or procedures stipulated in the study protocol.
9. Patient deprived of liberty or under legal protection (guardianship, legal protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, defined as the ratio of the number of refractory patients with an IBI score > 0 to the number of refractory patients. | 12 months for each patient
Specificity, defined as the ratio of the number of non-refractory patients with an IBI score = 0 to the number of non-refractory patients. | 12 months for each patient

SECONDARY OUTCOMES:
The sensitivity of the IBI score will be presented at different measurement times in a similar way to the primary endpoint. | 36 months for each patient
The specificity of the IBI score will be presented at different measurement times in a similar way to the primary endpoint. | 36 months for each patient
Clinico-pathological parameters will be presented by group (IBI score=0 vs >0) using standard descriptive statistics. | 36 months for each patient
Imaging parameters will be presented by group (IBI score=0 vs >0) using standard descriptive statistics. | 36 months for each patient
Progression-free survival (PFS) rates (time from inclusion to progression or death from any cause) will be estimated with their 95% confidence intervals using the Kaplan-Meier method. | 36 months for each patient

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Institut de Cancérologie de l'Ouest, Angers
  - CHU de Bordeaux, Bordeaux
  - Centre François Baclesse, Caen
  - CHU de Lille, Lille
  - CHU de Lyon, Lyon
  - Hôpital La Timone, Marseille
  - CHU Hôtel Dieu, Nantes
  - CHU de Poitiers, Poitiers
  - IUCT-O, Toulouse